CLINICAL TRIAL: NCT03861819
Title: Feasibility of Vigorous-Intensity Interval Training in Adults With Nonalcoholic Steatohepatitis
Brief Title: Feasibility of VIIT in Adults With NASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00087286
Record Dates: First submitted 2019-02-12; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Nonalcoholic Steatohepatitis (NASH); Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis; Liver Diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VIIT Intervention (Experimental): This is a single-arm trial. The intervention itself proceeds as follows: After approximately 5 minutes of warmup subjects will perform 10 intervals of VIIT: 30 seconds of vigorous intensity exercise followed by 60 seconds of rest. Rated Perceived Exertion (RPE) will be rated by 15-point Borg scale; should correspond to HR/10 at end of each interval. The subject will self-adjust the intensity of the exercise bouts and will be encouraged by the researcher to achieve the desired intensity. The exercise session will finish with a short cool-down period and will last no more than 25 minutes in total.
  Interventions: Behavioral: Vigorous-intensity interval training (VIIT)

INTERVENTIONS:
Behavioral: Vigorous-intensity interval training (VIIT) — Subjects will be fitted with a heart rate monitor around the chest and a baseline 4ml blood sample will be drawn. Vigorous intensity interval training will correspond to heart rate (HR) range of 80-90% of heart rate at age-predicted heart rate maximum (220-age). After approximately 5 minutes of warmup subjects will perform 10 intervals of VIIT: 30 seconds of vigorous intensity exercise followed by 60 seconds of rest. Rated Perceived Exertion (RPE) will be rated by 15-point Borg scale; should correspond to HR/10 at end of each interval. The subject will self-adjust the intensity of the exercise bouts and will be encouraged by the researcher to achieve the desired intensity. The exercise session will finish with a short cool-down period and will last no more than 25 minutes in total. A 4ml blood sample will be drawn immediately following the exercise session and 2-hours after exercise cessation.

SUMMARY:
The purpose of this study is to determine whether patients with stage 1-3 NASH-related fibrosis are able to complete a single vigorous-intensity interval training (VIIT) session on an indoor rowing machine and provide blood samples before and afterwards. The results of this study will provide the foundation for future research on the role of VIIT in treating NASH.

DETAILED DESCRIPTION:
Background & Significance:

The increasing prevalence of obesity and diabetes has prompted a global epidemic of nonalcoholic fatty liver disease affecting 15-30% of the general population. Of those with nonalcoholic fatty liver disease, 25% develop NASH and are at increased risk for progressive hepatic fibrosis and cirrhosis. NASH-related cirrhosis is now the second leading indication of liver transplantation in the United States. For the treatment of NASH, life-style modification with diet and exercise is mandatory. Diet and exercise-induced weight loss >5% total body weight improves NASH and reverses hepatic fibrosis, the primary determinant of liver related morbidity and mortality. While weight loss has remained fundamental to disease management it is mistaken as the only assessment for exercise-mediated improvements in NASH. Exercise alone has been shown to improve NASH irrespective of weight loss; however, how exercise works is unclear. Defining an understanding of how exercise effectively treats NASH is an urgent and unmet need that will optimize exercise prescriptions and facilitate identifying candidate therapeutic targets that mimic exercise response for those patients unable to sustain life-style modifications.

One potential mechanism for exercise improving NASH is through skeletal muscles' signaling proteins, known collectively as myokines. During exercise, myokines are released from skeletal muscle into the circulation where they communicate with several organs, including the liver. Emerging evidence suggests that myokines - particularly myokine interleukin 6 (IL-6) -directly regulates liver interleukin (IL)-8.

Our preliminary data demonstrates that in NASH patients, serum IL-8 is independently associated with hepatic fibrosis and differentially expressed by fibrotic stage. Whether exercise-mediated myokine IL-6 improves NASH-related fibrosis through reductions in IL-8 remains a gap in knowledge.

Myokine IL-6 release into the circulation has been shown to be dependent on the amount of skeletal muscle involved during exercise and level of exercise intensity. Thus, full-body movements performed at high-intensity may release the greatest amounts of myokine IL-6. Vigorous-intensity interval training (VIIT) has not been tested in patients with NASH. Additionally, VIIT in NAFLD has been traditionally performed on a cycle ergometer or treadmill, which greatly limits maximal skeletal muscle utilization during exercise. Since myokine release from skeletal muscle is hypothesized as a critical mechanism of exercise-mediated benefits in NAFLD, the investigators are proposing conducting a feasibility study of a single VIIT session in patients with NASH using an indoor rower. To measure IL-6 myokine response and subsequent changes in serum IL-8 the investigators will collect blood samples prior, immediately after, and 2-hours following a single VIIT session.

Design & Procedures:

12 adults, 18-59 yrs. of age, with NASH-related fibrosis (stage 1-3) will undergo a single VIIT session where blood will be collected prior, immediately following, and 2-hours after exercise:

* Visit 1: The initial visit will take place at the Duke Hepatology Clinic by Dr. Oliver Glass, PhD and Dr. Manal Abdelmalek MD MPH, and will last approximately 30 minutes. We will explain the study and consent form in detail and on an individual basis, and participants will have the opportunity to take the consent home and consider it. If a potential subject decides to consent during this visit, participants will be scheduled for visits 2 and 3. If a potential subject needs more time to consider the consent, participants will have a phone number to call to let study staff know that they wish to move forward with visits 2 and 3, and participants will be consented in person at visit 2 before any study activities take place.
* Visit 2: This 1-hour visit will take place at the Duke Integrative Medicine. Participants will be instructed on proper form and biomechanics of exercising on an indoor rowing machine. This session will ensure subjects are able to perform indoor rowing properly and safely.
* Visit 3: Subjects will be fitted with a heart rate monitor around the chest and a baseline 4ml blood sample will be drawn. Vigorous intensity interval training will correspond to heart rate (HR) range of 80-90% of heart rate at age-predicted heart rate maximum (220-age). After approximately 5 minutes of warmup subjects will perform 10 intervals of VIIT: 30 seconds of vigorous intensity exercise followed by 60 seconds of rest. Rated Perceived Exertion (RPE) will be rated by 15-point Borg scale; should correspond to HR/10 at end of each interval. The subject will self-adjust the intensity of the exercise bouts and will be encouraged by the researcher to achieve the desired intensity. The exercise session will finish with a short cool-down period and will last no more than 25 minutes in total. A 4ml blood sample will be drawn immediately following the exercise session and 2-hours after exercise cessation.

Participants may opt-in/opt-out of the option to have their blood samples stored for future research on whether acute exercise alters other myokines besides IL-6 and IL-8. Additionally, future research would evaluate whether acute exercise changes other immune-inflammatory blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-59
* Histologically confirmed nonalcoholic steatohepatitis and fibrosis (stage 1-3) from liver biopsy
* Able to row on an indoor rowing apparatus
* Not participating in regular physical exercise (more than 60 minutes of moderate intensity or 30 minutes of vigorous intensity exercise per week)
* Not actively trying to lose weight through a dietary approach
* No absolute contra-indications to exercise: recent (<6 months) acute cardiac event unstable angina, uncontrolled dysrhythmias causing symptoms or hemodynamic compromise, symptomatic aortic stenosis, uncontrolled symptomatic heart failure, acute pulmonary embolus, acute myocarditis or pericarditis, suspected or known dissecting aneurism and acute systemic infection
* No other form of chronic liver disease (as confirmed by serology and histology)
* No liver cirrhosis (stage 4 fibrosis on liver biopsy) or a clinical diagnosis of cirrhosis as ascertained by a hepatologist
* No coronary artery disease or chronic obstructive pulmonary disease.
* No diagnosis of malignancy (except non-melanoma skin cancer)
* No past or present history of portal hypertension (esophageal varices, ascites, hepatic encephalopathy)
* No use of immunosuppression or chronic nonsteroidal anti-inflammatory medication
* No more than 14 drinks per week (if male) or 7 drinks a week (if female) in the last 2 years
* Cognitively able to provide consent
* Able to read, write, and understand English
* Transportation to the exercise and testing facility

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by adherence to the intervention. | Feasibility will be assessed after all subjects have completed the study, after a 12-month recruiting period.
  This study is designed to assess the feasibility of a VIIT intervention for adults with NASH-related fibrosis. Adherence will be measured as the % of subjects who are able to achieve the protocol target of 80% of their max heart rate during the intervention.
Feasibility as measured by ease of recruiting | Feasibility will be assessed after all subjects have completed the study, after a 12-month recruiting period.
  This study is designed to assess the feasibility of a VIIT intervention for adults with NASH-related fibrosis. Ease of recruiting will be determined by assessing whether the accrual target was met within the 12-month recruitment timeline.

SECONDARY OUTCOMES:
Change in myokine response | Secondary outcome measures will be assessed immediately post-exercise and 2-hours following exercise.
  The secondary outcome will be the change is 1L-6 and IL-8 cytokine response before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Integrative Medicine, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided